CLINICAL TRIAL: NCT05236309
Title: Taipei City Hospital Linsen Chinese Medicine and Kunming Branch
Brief Title: Investigation on the Epidemic Prevention Effect of Using Chinese Medicine During the Severe Acute Respiratory Syndrome Coronavirus 2 (SARS-CoV-2) Outbreak.
Status: Completed | Type: Observational
Sponsor: Taipei City Hospital (Other Government)
Responsible Party: Principal Investigator, Chung-Hua Hsu, Clinical Professor, Taipei City Hospital
Other Study IDs: TCHIRB-11009019-E
Record Dates: First submitted 2021-11-18; First posted 2022-02-11 (Actual); Last update posted 2022-03-02 (Actual); Status verified 2022-02

CONDITIONS: COVID-19 Pandemic
Keywords: Chinese medicine
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- JGF (Jing-Guan-Fang): Traditional Chinese Medicine Decoction: JGF group: 100ml JGF decoction per day at least 1 week
  Interventions: Drug: Jing-Guan-Fang(JGF) : Chinese herbal decoction
- NO JGF: NO JGF group: None use traditional Chinese medicine(JGF)

INTERVENTIONS:
Drug: Jing-Guan-Fang(JGF) : Chinese herbal decoction — Use 100ml JGF decoction per day as a preventive measure for patients with COVID-19.
  Other Names: Chinese herbal decoction
  Groups: JGF (Jing-Guan-Fang): Traditional Chinese Medicine Decoction

SUMMARY:
Taking a regional hospital as an example, the investigators will discuss the changes in the community cumulative incidence rate(CIR) and the epidemic prevention effect of using Chinese medicine during the SARS-CoV-2 outbreak.

Main purpose:

Retrospective case study to explore the effect of traditional Chinese medicine on the prevention of SARS-CoV-2.

Secondary purpose:

If there are related side effects after taking Chinese medicine.

DETAILED DESCRIPTION:
The large-scale coronavirus epidemic is a major global public health challenge in the 21st century. Since the 2003 Severe acute respiratory syndrome (SARS) epidemic spread globally and caused hundreds of deaths, the Middle East respiratory syndrome (Middle East respiratory syndrome, MERS) and coronavirus disease 2019(COVID-19) has caused a large-scale global spread and also caused a huge impact on the public health and medical system. In the country's current epidemic (Aug 1, 2021), more than 15,000 people have been diagnosed, and the number of deaths has exceeded 800. Among them, the Taipei epidemic is the most severe, and the Wanhua District of Taipei City is the hot zone. The investigators will discuss the changes in accumulation incidence rate(CIR) of the community and the epidemic prevention effect of using Chinese medicine during the SARS-CoV-2 outbreak.

This is a retrospective case study to explore the effect of traditional Chinese medicine on the prevention of SARS-CoV-2 and discuss if there are related side effects after taking Chinese medicine.

ELIGIBILITY:
Inclusion Criteria:

- From January 1, 2020 to July 31, 2021, Chinese medicine is used for patients with new coronary pneumonia epidemic prevention.

Exclusion Criteria:

1. Patients who do not use traditional Chinese medicine for the prevention of new coronary pneumonia.
2. Patients who have signed and refused to provide medical records.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The subjects of this study are patients who went to the Taipei City Hospital Linsen Chinese Medicine and Kunming Branch from January 1, 2020, to July 31, 2021. It is estimated that the medical records of 1,000 patients who use traditional Chinese medicine for new coronary pneumonia prevention and control will be collected as the experimental group, and they will be randomly matched. The medical records of 1,000 patients who have not used Chinese medicine as a control group for the prevention of new coronary pneumonia, a total of 2,000.
Sampling Method: Probability Sample
Enrollment: 2000 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2021-07-31 (Actual); Study Completion 2021-11-18 (Actual)

PRIMARY OUTCOMES:
Investigation on the effect of using traditional Chinese medicine to prevent SARS-CoV-2 infection in two groups with cumulative incidence rate(CIR). | 18 months
  Compare the dangerous states within two groups with CIR.

CONTACTS AND LOCATIONS:
Locations (1):
- Taipei City Hospital, Taipei, Taiwan